CLINICAL TRIAL: NCT02573285
Title: Simple Aspiration for Initial Management of Primary Spontaneous Pneumothorax in Children: A Multi-Center Pilot Study
Brief Title: Spontaneous Pneumothorax in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other); Indiana University (Other); Medical College of Wisconsin (Other); Northwestern University (Other); Nationwide Children's Hospital (Other); University of Chicago (Other); University of Louisville (Other); University of Michigan (Other); Washington University School of Medicine (Other); Children's Mercy Hospital Kansas City (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-1188; A539790 (Other: UW, Madison); SMPH/SURGERY (Other: UW, Madison)
Record Dates: First submitted 2015-10-05; First posted 2015-10-09 (Estimated); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Spontaneous Pneumothorax
MeSH Terms: conditions — Pneumothorax | interventions — Thoracentesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simple Aspiration (Active Comparator): Subjects in this arm will undergo initial management of their pneumothorax with a simple aspiration procedure. The procedure will involve placement of a small catheter into the chest cavity and applying negative pressure to manually aspirate the air out of the chest cavity, which will allow the lung to re-expand.
  Interventions: Procedure: Simple Aspiration
- Surgeon Preference (Active Comparator): Subjects that choose the surgeon preference arm of the study are enrolling for prospective data collection only. These subjects will not have any portion their care directed by the study protocol. The decision to proceed with any treatment or intervention will be made jointly by the surgeon and the patient and his or her legal guardian. Any standard treatment option may be utilized, including simple aspiration, chest tube placement, or an operation (VATS).
  Interventions: Procedure: Surgeon Preference

INTERVENTIONS:
Procedure: Simple Aspiration — Aspiration of pneumothorax with a small-bore catheter
  Other Names: Thoracentesis
  Arms: Simple Aspiration
Procedure: Surgeon Preference — Any standard treatment option may be utilized for the treatment of the pneumothorax, including simple aspiration, chest tube placement, or an operation (VATS).
  Arms: Surgeon Preference

SUMMARY:
The objective of this multi-center, non-randomized, prospective pilot study is to examine the rate of successful primary spontaneous pneumothorax (PSP) resolution using the simple aspiration technique.

In this study, eligible subjects diagnosed with PSP at eleven participating large children's hospitals (members of the Midwest Pediatric Surgical Clinical Research Consortium) will be enrolled and offered a choice of management with either the simple aspiration protocol or management according to their surgeon's preference, which may include simple aspiration, chest tube placement, or rarely, an operation.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, multi-center pilot study involving children (age 12-17 years old) who present with a first episode of primary spontaneous pneumothorax (PSP) that requires treatment. Treatment with simple aspiration has been researched in adults but it has not been investigated in children. For this reason, this will be a pilot study design with two non-randomized groups. Since some pediatric surgeons have started to offer this treatment in children and some of the adult studies include adolescent patients, simple aspiration is considered a standard of care treatment at many institutions, and is performed as part of standard care at UW. Patient and Provider communication regarding treatment options and the Patient and Provider choice choice of treatment play a large role both in the standard of care for PSP and this research study.

Potential subjects will be identified by a consulting surgeon (who will be a study team member as all pediatric surgeons are on this application) when surgical consultation is requested for acute management of a child with spontaneous pneumothorax. This most commonly occurs in the emergency department after a chest X-ray is obtained as part of the usual evaluation for the associated symptoms of pain and shortness of breath. Medical records may be reviewed to confirm eligibility prior to approaching potential subjects and their parents/guardians for assent/consent. The consulting surgeon will also assess patient eligibility by screening for inclusion and exclusion criteria. If all eligibility criteria are met, the consulting surgeon will notify a member of the study staff about the potential subject.

A member of the research team will explain the study rationale and procedures in detail with potential subjects and their legal guardian upon surgical consultation. All written information will be reviewed and all questions answered. A study physician will be available at all times for any consent-related questions. The potential subject and legal guardian will have up to one hour to consider if they would like to participate in the study. The child's legal guardian will sign the informed consent, and the subject will sign assent.

Once consent/assent is obtained subjects and their parents/guardians will have the choice of consenting to initial management with either the simple aspiration protocol (aspiration group) or according to the preferences of the treating surgeon (preference group). All patients will be properly informed of the options for each arm during the consent discussion, most of the information is conveyed during the clinical treatment discussion with the patients which is then incorporated into the consent discussion. Patient preference and choice of treatment plays a large role in the standard of care methods for treating PSP and subject preference and choice will play just as strong a role in this research study.

As a pilot study, we aim to enroll 32 subjects in the aspiration arm across all participating institutions and 48 subjects will enroll into the preference arm. Since all medical treatments performed during the study are considered standard of care, the only research components of this study include the subject's self-allocation to a particular study arm (even though patient choice is just as strong a role in standard of care, there are defined arms for this research study) and the recording of medical and billing data for each subject, as well as a follow-up phone call to the subject.

Aspiration Arm:

Subjects in this arm will undergo initial management of their pneumothorax with a simple aspiration procedure according to standard care described here. The procedure will involve placement of a small catheter into the chest cavity and applying negative pressure to manually aspirate the air out of the chest cavity, which will allow the lung to re-expand. The aspiration catheter will be less than or equal to 12 French in diameter. Further details of the type of device and size of catheter will be determined by the surgeon and will depend on the devices available for standard practice at each participating institution. The procedure may be performed with local anesthetic, with or without sedation, depending on surgeon judgment and available resources or standard practice at each participating institution. The procedure may be performed with or without image guidance (i.e. ultrasound or fluoroscopy) during the aspiration, but a chest X-ray must be obtained at the conclusion of the procedure, with the catheter still in place, to verify successful expansion of the lung and for comparison with subsequent chest X-rays. A small residual pneumothorax after the initial aspiration procedure may still be deemed a success. Successful aspiration at the time of the initial aspiration procedure will be defined as: expansion of the lung apex to the top of the 4th rib or higher and expansion at the lateral chest wall to the 6th rib or higher. A failure will be defined as a residual pneumothorax that is not limited to the apex and extends laterally down the chest wall below the 6th rib. If the first post-procedure chest X-ray demonstrates failure of adequate lung expansion, the existing catheter may be used for one additional aspiration attempt, with application of negative pressure followed by another chest X-ray.

After the aspiration procedure, the subject will be admitted to the hospital for a minimum observation period of 6 hours. The small catheter will be capped and left in place and the insertion site covered by an occlusive dressing, such that this same catheter could be utilized in the event of failure of the aspiration procedure. After 6 hours, a second chest X-ray will be obtained to assess for recurrent pneumothorax or enlargement of a small residual pneumothorax. If the pneumothorax is stable or smaller in size after 6 hours of observation, then the catheter will be removed and the patient discharged to home. However, if the pneumothorax recurs or enlarges after 6 hours, then the aspiration procedure has failed. The existing catheter could be uncapped and used as an indwelling chest tube for a more prolonged period of chest drainage, but all management is according to the surgeon's preference and standard practice. At any time, if the aspiration procedure is determined to be a failure, by either inadequate lung expansion or recurrent pneumothorax, the patient will be managed according to the judgment and standard practice of the treating surgeon.

Preference Arm:

Subjects that choose the surgeon preference arm of the study are enrolling for prospective data collection only. These subjects will not have any portion their care directed by the study protocol. The decision to proceed with any treatment or intervention will be made jointly by the surgeon and the patient and his or her legal guardian. Any standard treatment option may be utilized, including simple aspiration, chest tube placement, or an operation, video-assisted thoracoscopic surgery (VATS). If the surgeon's preference and standard treatment is simple aspiration but the patient does not want the aspiration procedure, then the surgeon will perform an alternative treatment option, such as chest tube placement or VATS.

Management strategies in the preference group may include placement of an indwelling chest tube, with or without thoracoscopic resection of blebs (VATS), and may also include a simple aspiration procedure if recommended by the treating surgeon.

For both arms, a telephone survey will be conducted at approximately one year from enrollment. The primary purpose is to ascertain whether the subject has sought additional medical treatment at another facility for unresolved or recurrent pneumothorax and time to recurrence. Additionally, we wish to know if the subject has ongoing or intermittent episodes of symptoms attributed to pneumothorax for which he/she has not sought medical treatment. A yearly chart audit will continue for 5 additional years to determine if any further treatment was needed for the initial pneumothorax.

ELIGIBILITY:
Inclusion Criteria:

Each subject must meet all of the following inclusion criteria to be enrolled in the study:

1. Age greater than or equal to 12 years and less than 18 years at date of enrollment.
2. First time seeking medical attention for symptoms related to primary spontaneous pneumothorax.
3. Consulting surgeon determines that intervention is required for treatment of spontaneous pneumothorax.

Exclusion Criteria:

1. Patients with a previous episode of pneumothorax on the same side of the chest that required medical treatment in the past.
2. Pneumothorax is secondary to a co-morbid medical condition (underlying pulmonary disease, malignancy, or trauma).
3. Pneumothorax is small and amenable to observation: size <2cm space between lung and chest wall at the apex and clinically stable patient with minimal symptoms.
4. Bilateral pneumothorax.
5. Unstable patient in need of emergent intervention at surgeon discretion.
6. Patients who are known to be pregnant.
7. Patients in the custody of the state.
8. Patients who are currently prisoners.
9. Non-English speaking.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2016-03-10 (Actual); Primary Completion 2018-06-04 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
The success rate of simple aspiration of initial management of primary spontaneous pneumothorax in children | At the time of post-procedure chest X-ray
  Adequate expansion of the lung without the need for additional intervention from admission until discharge for PSP

SECONDARY OUTCOMES:
Rate of recurrent pneumothorax | After 6 hours of observation from treatment to 1 year
  Number of recurrent pneumothoraces
Time to recurrence of pneumothorax | From initial treatment up one year
  Recurrence of a pneumothorax within 1 year of initial hospitalization for pneumothorax
Total length of hospital stay | Up to 7 days
  Time between admission until discharge for treatment of pneumothorax
Need for operative intervention (VATS) following initial management | Up to 1 year
  Surgical intervention needed for pneumothorax (yes/no)
Number of chest X-rays and/or CT scans | Up to 7 days
  Count of the number of chest X-rays completed or CT scans completed for pneumothorax
Procedural complications | Up to 7 days
  Count of the number of complications during the initial hospitalization for pneumothorax
Total aggregate hospital costs for initial hospitalization | Up to 7 days
  Aggregate hospital charges during initial admission for pneumothorax
Need for further intervention for spontaneous pneumothorax | Between 1 year and 5 year follow-up
  Treatment or intervention needed for spontaneous pneumothorax after the 1 year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Charles Leys, MD, MSCI, Principal Investigator — Pediatric Surgeon, American Family Children's Hospital
Locations (1):
- American Family Children's Hospital, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
No sharing

REFERENCES:
- [Result] Baumann MH, Strange C, Heffner JE, Light R, Kirby TJ, Klein J, Luketich JD, Panacek EA, Sahn SA; AACP Pneumothorax Consensus Group. Management of spontaneous pneumothorax: an American College of Chest Physicians Delphi consensus statement. Chest. 2001 Feb;119(2):590-602. doi: 10.1378/chest.119.2.590. PMID 11171742
- [Result] MacDuff A, Arnold A, Harvey J; BTS Pleural Disease Guideline Group. Management of spontaneous pneumothorax: British Thoracic Society Pleural Disease Guideline 2010. Thorax. 2010 Aug;65 Suppl 2:ii18-31. doi: 10.1136/thx.2010.136986. No abstract available. PMID 20696690
- [Result] Noppen M, Alexander P, Driesen P, Slabbynck H, Verstraeten A. Manual aspiration versus chest tube drainage in first episodes of primary spontaneous pneumothorax: a multicenter, prospective, randomized pilot study. Am J Respir Crit Care Med. 2002 May 1;165(9):1240-4. doi: 10.1164/rccm.200111-078OC. PMID 11991872
- [Result] Robinson PD, Cooper P, Ranganathan SC. Evidence-based management of paediatric primary spontaneous pneumothorax. Paediatr Respir Rev. 2009 Sep;10(3):110-7; quiz 117. doi: 10.1016/j.prrv.2008.12.003. Epub 2009 May 21. PMID 19651381
- [Result] Sahn SA, Heffner JE. Spontaneous pneumothorax. N Engl J Med. 2000 Mar 23;342(12):868-74. doi: 10.1056/NEJM200003233421207. No abstract available. PMID 10727592
- [Result] Gupta D, Hansell A, Nichols T, Duong T, Ayres JG, Strachan D. Epidemiology of pneumothorax in England. Thorax. 2000 Aug;55(8):666-71. doi: 10.1136/thorax.55.8.666. PMID 10899243
- [Result] Wakai A, O'Sullivan RG, McCabe G. Simple aspiration versus intercostal tube drainage for primary spontaneous pneumothorax in adults. Cochrane Database Syst Rev. 2007 Jan 24;(1):CD004479. doi: 10.1002/14651858.CD004479.pub2. PMID 17253510